CLINICAL TRIAL: NCT03423186
Title: An Open, Non-controlled, Parallel, Ascending Multiple-dose, Multicenter Study to Assess Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of SOBI003 in Pediatric MPS IIIA Patients
Brief Title: A Study to Assess the Safety and Tolerability of SOBI003 in Pediatric MPS IIIA Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOBI003-001
Record Dates: First submitted 2018-01-29; First posted 2018-02-06 (Actual); Results first posted 2021-04-22 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Sanfilippo Syndrome Type A (MPS IIIA)
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Intervention Model Description: The study was designed to include three arms, up to 20 mg/kg. After a company decision to end the development of the compound it was decided to not start a third cohort, but if stated safe the dose could increase up to 20 mg/kg in cohort 1 and 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose group 1 (Experimental): SOBI003 dose 3 mg/kg once weekly for 24 weeks
  Interventions: Drug: SOBI003
- Dose group 2 (Experimental): SOBI003 dose 10 mg/kg once weekly for 24 weeks
  Interventions: Drug: SOBI003

INTERVENTIONS:
Drug: SOBI003 — Weekly i.v.infusion
  Other Names: Modified recombinant human sulphamidase

SUMMARY:
MPS IIIA, also known as Sanfilippo A, is an inherited lysosomal storage disease (LSD). MPS IIIA is caused by a deficiency in sulfamidase, one of the enzymes involved in the lysosomal degradation of the glycosaminoglycan (GAG) heparan sulfate (HS). The natural course of MPS IIIA is characterized by devastating neurodegeneration with initially mild somatic involvement. The aims of the present study is to assess the dose related safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of SOBI003, a chemically modified recombinant human (rh) Sulfamidase developed as an enzyme replacement therapy (ERT).

DETAILED DESCRIPTION:
This is an open-label, non-controlled, parallel, sequential ascending multiple-dose, multicenter study to assess the dose related safety, tolerability, PK and PD of SOBI003 in pediatric MPS IIIA patients. Patients between 1 and 6 years of age who have not received previous treatment for MPS IIIA with an ERT, gene- or stem cell therapy will be eligible to participate in the study. The study is planned to consist of 3 dose cohorts, each comprising 3 patients. Treatment initiations will be staggered within each cohort in order to be able to observe, interpret and treat possible adverse reactions. SOBI003 is administered as weekly i.v. infusions over a period of 24 weeks. Upon completion of the 24-week treatment period with satisfactory tolerability, the patient is offered to receive continued SOBI003 treatment by participation in an extension study.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained from the patient's legally authorized representative(s)
2. Patients with MPS IIIA, as confirmed by both:

   * A documented deficiency in sulfamidase enzyme activity in concordance with a diagnosis of MPS IIIA, and
   * Normal enzyme activity level of at least one other sulfatase measured in leukocytes
3. Chronological age of ≥12 and ≤72 months (i.e., 1 to 6 years) at the time of the first SOBI003 infusion and a developmental age ≥12 months at screening as assessed by the Vineland Adaptive Behavior Scales, Second Edition (VABS-II)
4. Medically stable patient who is expected to be able to comply with study procedures

Exclusion Criteria:

1. At least one S298P mutation in the SGSH gene
2. Contraindications for anesthetic procedures, surgical procedure (venous access port) MRI scans and/or lumbar punctures
3. History of poorly controlled seizures
4. Patients is currently receiving psychotropic or other medications which in the investigator's opinion, would be likely to substantially confound test results
5. Significant non-MPS IIIA-related central nervous system (CNS) impairment or behavioral disturbances, which in the investigator's opinion, would confound the scientific integrity or interpretation of study assessments
6. Prior administration of stem cell or gene therapy, or ERT for MPS IIIA
7. Concurrent or prior (within 30 days of enrolment into this study) participation in a study involving invasive procedures

Ages: 12 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Harmatz, MD, Principal Investigator — Childrens's Hospital and Research Center Oakland
Locations (4):
- United States (2):
  - Childrens's Hospital and Research Center, Oakland, California
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- Gazi University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Undecided

REFERENCES:
- [Derived] Harmatz P, Muenzer J, Ezgu F, Dalen P, Huledal G, Lindqvist D, Gelius SS, Wiken M, Onnestam K, Broijersen A. Chemically modified recombinant human sulfamidase (SOBI003) in mucopolysaccharidosis IIIA patients: Results from an open, non-controlled, multicenter study. Mol Genet Metab. 2022 Aug;136(4):249-259. doi: 10.1016/j.ymgme.2022.06.008. Epub 2022 Jun 28. PMID 35835061

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Group 1 | Dose Group 2
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Group 1 | Dose Group 2 | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: months] — Age at day of first infusion (months)
  months | 46.3 (24.2) | 29.0 (12.2) | 37.7 (19.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by Adverse Events Frequencies (by Type and Severity)
Description: Number of adverse events, by type and severity, from start of infusion up to 24 weeks
Time Frame: From start of first infusion up to Week 24
Measure: Number; unit: number of events
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
number of events
  Any adverse event | 53 | 128
  Any non-treatment emergent serious adverse event | 0 | 1
  Any treatment emergent adverse event (TEAE) | 53 | 124
  Any drug-related TEAE | 27 | 74
  Any non-serious TEAE | 52 | 121
  Any serious TEAE | 1 | 3
  Any serious drug-related TEAE | 0 | 0
  Any TEAE leading to study and/or treatment withdrawal | 0 | 0
  Any drug-related TEAE leading to study and/or treatment withdrawal | 0 | 0
  Any serious TEAE leading to study and/or treatment withdrawal | 0 | 0
  Any TEAE leading to death | 0 | 0
  Any Infusion related Reaction | 17 | 27

2. Secondary Outcome: The Observed Serum Concentration Immediately Before the Start of Infusion of SOBI003
Description: The observed serum concentration immediately before the start of infusion of SOBI003 (CPre-dose).
Time Frame: Weeks 1, 2, 3, 4, 8, 12, and 24
Population: The table report number of available pharmacokinetic (PK) samples
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
ng/mL
  Week 1 | NA [NA to NA] — Levels below LLOQ | NA [NA to NA] — Levels below LLOQ
  Week 2 | 58.4 [33.0 to 62.2] | 109.0 [85.7 to 137.0]
  Week 3: number analyzed (Participants) | 2 | 2
  Week 3 | 68.85 [55.2 to 82.5] | 135.5 [114.0 to 157.0]
  Week 4 | 71.4 [NA to 97.7] — Levels below LLOQ | 49.8 [31.4 to 603.0]
  Week 8: number analyzed (Participants) | 3 | 2
  Week 8 | NA [NA to 27.0] — Levels below LLOQ | 25.5 [NA to 51] — Levels below LLOQ
  Week 12: number analyzed (Participants) | 2 | 3
  Week 12 | 33.75 [26.6 to 40.9] | NA [NA to 10.3] — Levels below LLOQ
  Week 24 | NA [NA to NA] — Levels below LLOQ | 16.4 [NA to 90.0] — Levels below LLOQ

3. Secondary Outcome: The Observed Serum Concentration at the End of Infusion of SOBI003
Description: The observed serum concentration at the end of infusion of SOBI003 (CEnd of inf)
Time Frame: Weeks 1, 2, 3, 4, 8, 12, and 24
Population: Number of analysed are available samples
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
ng/mL
  Week 1 | 33800 [29500 to 36400] | 87500 [75300 to 114000]
  Week 2: number analyzed (Participants) | 2 | 2
  Week 2 | 34950 [33300 to 36600] | 108200 [99400 to 117000]
  Week 3: number analyzed (Participants) | 2 | 2
  Week 3 | 36750 [31300 to 42200] | 82700 [73300 to 92100]
  Week 4 | 35700 [16150 to 36600] | 77400 [71800 to 102000]
  Week 8 | 20800 [65.5 to 36600] | 50900 [33300 to 68600]
  Week 12 | 30500 [32.5 to 36700] | 56900 [56100 to 71000]
  Week 24 | 17500 [47.5 to 35400] | 93500 [69700 to 103000]

4. Secondary Outcome: The Time of the End of the Infusion of SOBI003
Description: The time of the end of infusion of SOBI003 (tEnd of inf)
Time Frame: Weeks 1, 2, 3, 4, 8, 12, and 24
Population: Number of analysed are available samples
Measure: Median (Full Range); unit: Hours
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Hours
  Week 1 | 4.57 [4.27 to 4.62] | 4.33 [4.02 to 4.33]
  Week 2: number analyzed (Participants) | 2 | 2
  Week 2 | 4.565 [4.30 to 4.83] | 4.245 [4.07 to 4.42]
  Week 3: number analyzed (Participants) | 2 | 2
  Week 3 | 4.28 [4.13 to 4.43] | 4.1 [3.98 to 4.22]
  Week 4 | 4.28 [4.05 to 4.50] | 4.42 [4.27 to 4.90]
  Week 8: number analyzed (Participants) | 3 | 2
  Week 8 | 4.85 [4.42 to 6.58] | 8.17 [8.17 to 8.17]
  Week 12 | 4.23 [4.10 to 6.42] | 6.83 [5.08 to 7.03]
  Week 24 | 4.45 [4.08 to 4.53] | 4.75 [4.47 to 5.57]

5. Secondary Outcome: The Maximum Observed Serum Concentration of SOBI003
Description: The Maximum Observed Serum Concentration of SOBI003 (Cmax)
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose on Weeks 1, 4, 12, and 24
Population: Samples was taken centrally and/or peripherally.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
ng/mL
  Week 1 | 33800 [29500 to 36400] | 87500 [75300 to 114000]
  Week 4 | 35700 [16150 to 36600] | 77400 [71800 to 102000]
  Week 12 | 20800 [65.5 to 36400] | 56900 [56100 to 71000]
  Week 24 | 17500 [47.5 to 35400] | 93500 [69700 to 103000]

6. Secondary Outcome: The Time at Which the Maximum Serum Concentration of SOBI003 is Observed
Description: The time after start of infusion at which the maximum serum concentration is observed (tmax)
Time Frame: Weeks 1, 4, 12, and 24
Measure: Median (Full Range); unit: Hours
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Hours
  Week 1 | 4.57 [4.27 to 4.62] | 4.33 [4.02 to 4.33]
  Week 4 | 4.28 [4.05 to 4.50] | 4.42 [4.27 to 4.90]
  Week 12 | 4.23 [4.10 to 6.42] | 6.83 [5.08 to 7.03]
  Week 24 | 4.45 [4.08 to 4.53] | 4.75 [4.47 to 5.57]

7. Secondary Outcome: The Minimum Observed Serum Concentration of SOBI003
Description: The minimum observed serum concentration of SOBI003 (CTrough)
Time Frame: Weeks 1, 4, 12, and 24
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
ng/mL
  Week 1 | NA [NA to 2010] — Levels below LLOQ | NA [NA to NA] — Levels below LLOQ
  Week 4 | 28.9 [NA to 61.3] — Levels below LLOQ | 115 [20.8 to 7730]
  Week 12 | 26.2 [17.0 to 32.5] | NA [NA to 29.7] — Levels below LLOQ
  Week 24 | 44.8 [NA to 47.5] — Levels below LLOQ | NA [14.6 to 9010] — Levels below LLOQ

8. Secondary Outcome: Clearance
Description: Clearance (CL) of SOBI003
Time Frame: Weeks 1, 4, 12, and 24
Measure: Median (Full Range); unit: (mL/h)/kg
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 2 | 2
(mL/h)/kg
  Week 1 | 10.4 [9.7 to 11.1] | 12.8 [12.0 to 13.6]
  Week 4 | 8.1 [8.0 to 8.2] | 12.75 [12.4 to 13.1]
  Week 12 | 9.5 [7.8 to 11.2] | 13.45 [12.1 to 14.8]
  Week 24 | 19.5 [10.2 to 28.8] | 10.4 [9.9 to 10.9]

9. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to 168 Hours
Description: Area under the serum concentration-time curve from time 0 to 168 hours (AUC 0-168h)
Time Frame: 0,1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168 hours post-dose on Weeks 1, 4,12, and 24
Population: Number of analysed are available samples
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
h*ng/mL
  Week 1: number analyzed (Participants) | 2 | 3
  Week 1 | 290044.5 [275152 to 304937] | 834411 [737687 to 2492658]
  Week 4: number analyzed (Participants) | 2 | 2
  Week 4 | 369915.5 [365435 to 374396] | 789106.5 [761760 to 816453]
  Week 12: number analyzed (Participants) | 2 | 2
  Week 12 | 324999.5 [267722 to 382277] | 749864 [674188 to 828540]
  Week 24: number analyzed (Participants) | 2 | 2
  Week 24 | 198973 [104009 to 293937] | 961516.5 [915941 to 1007092]

10. Secondary Outcome: The Half-life
Description: The half-life of SOBI003 in serum (T1/2)
Time Frame: Weeks 1, 4, 12, and 24
Measure: Median (Full Range); unit: Hours
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 2 | 2
Hours
  Week 1 | 19.8 [5.4 to 34.2] | 22.75 [5.8 to 39.7]
  Week 4 | 34.3 [29.7 to 38.9] | 7.65 [6.3 to 9.0]
  Week 12 | 40.95 [34.4 to 47.5] | 10.75 [8.8 to 12.7]
  Week 24 | 20.85 [9.3 to 32.4] | 15.95 [6.0 to 25.9]

11. Secondary Outcome: SOBI003 Concentration in Cerebrospinal Fluid
Description: SOBI003 concentration in cerebrospinal fluid
Time Frame: Weeks 12 and 24
Population: Number of analysed are available samples
Measure: Median (Full Range); unit: mg/L
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
mg/L
  Week 12: number analyzed (Participants) | 3 | 1
  Week 12 | NA [NA to NA] — Levels below LLOQ | 17.8 [17.8 to 17.8]
  Week 24 | NA [NA to NA] — Levels below LLOQ | 47.2 [12.2 to 64.6]

12. Secondary Outcome: Number of Patients Having Anti-drug Antibodies in Serum
Description: Number of patients in each dose group having anti-drug antibodies in serum
Time Frame: Weeks 2,4,8,12 and 24
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Participants
  Weeks 2 | 1 | 1
  Weeks 4 | 2 | 3
  Weeks 8 | 3 | 3
  Weeks 12 | 3 | 3
  Weeks 24 | 3 | 3

13. Secondary Outcome: Patients Having Anti-drug Antibodies in Cerebrospinal Fluid
Description: Percent of patients having anti-drug antibodies in cerebrospinal fluid
Time Frame: Weeks 12 and 24
Measure: Number; unit: percent of participants in dose group
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
percent of participants in dose group
  Week 12 | 33.3 | 66.7
  Week 24 | 66.7 | 100

14. Secondary Outcome: Change From Baseline in Heparan Sulfate Levels in Cerebrospinal Fluid
Description: Change from baseline, in percent, of Heparan Sulfate levels in cerebrospinal fluid
Time Frame: Baseline, weeks 12, and 24
Measure: Median (Full Range); unit: percent change
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
percent change
  Week 12 | -5.4 [-33.0 to 7.7] | -52.8 [-64.6 to -28.4]
  Week 24 | -17.5 [-26.5 to -14.7] | -50.9 [-59.4 to -21.2]

15. Secondary Outcome: Change From Baseline in Heparan Sulfate Levels in Serum
Description: Change from baseline in Heparan sulfate levels in serum
Time Frame: Weeks 2, 3, 4, 8, 12 and 24
Measure: Median (Full Range); unit: mg/L
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
mg/L
  Week 2 | -1.8070 [-1.891 to -0.660] | -1.7460 [-3.409 to -1.705]
  Week 3 | -1.22 [-2.006 to -0.220] | -1.9190 [-3.576 to -1.856]
  Week 4 | -1.9040 [-2.083 to -1.850] | -1.9229 [-3.770 to -1.268]
  Week 8 | -2.1030 [-2.210 to -1.615] | -1.8290 [-3.730 to -1.772]
  Week 12 | -1.8170 [-2.131 to -1.597] | -1.8340 [-3.729 to -1.722]
  Week 24 | -1.7480 [-2.207 to -1.657] | -1.8310 [-3.722 to -1.818]

16. Secondary Outcome: Change From Baseline in Heparan Sulfate Levels in Urine
Description: Change from baseline in Heparan sulfate levels in urine
Time Frame: Weeks 2, 3, 4, 8, 12 and 24
Measure: Median (Full Range); unit: g/mol
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
g/mol
  Weeks 2 | -456.2 [-496.1 to -298] | -561.1 [-592.1 to -231.9]
  Weeks 3 | -494.67 [-592.1 to -390.0] | -597.4 [-618.8 to -309.3]
  Weeks 4 | -498.53 [-575.8 to -422.79] | -503.465 [-672.17 to -334.76]
  Weeks 8 | -474.7 [-542.22 to -460.95] | -666.81 [-672.42 to -341.70]
  Weeks 12 | -534.1 [-540.71 to -442.33] | -640.2 [-668.83 to -326.13]
  Weeks 24 | -421.98 [-557.33 to -258.1] | -695.9 [-698.03 to -348.05]

17. Secondary Outcome: Change From Baseline in Neurocognitive Development Quotient
Description: Quotient between age equivalent score and age, 0 - 100%, where high values are desirable. The age equivalent score represent the age of the typical and normal individual who would achieve the same result as the one who was tested.
  The age equivalent scores are assessed by the Bayley Scales of Infant and Toddler Development®, third edition cognitive subtest or the Kaufman Assessment Battery for Children, Second edition.
  The Bayley Scales of Infant and Toddler Development-Third Edition is an individually administered test designed to assess developmental functioning of infants and toddlers. The Bayley-III assesses development in five areas: cognitive, language, motor, social-emotional, and adaptive behavior.
  The Kaufman Assessment Battery for Children (K-ABC) is a clinical instrument for assessing cognitive development.
Time Frame: Week 24
Measure: Median (Full Range); unit: unitless
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
unitless | -8.7 [-11.2 to -4.9] | -15.68 [-53.3 to 4.1]

18. Secondary Outcome: Change From Baseline in Age-equivalence Score
Description: The age equivalent score represent the age in months of the typical and normal individual who would achieve the same result as the one who was tested.
  The age equivalent scores are assessed by the Bayley Scales of Infant and Toddler Development®, third edition cognitive subtest or the Kaufman Assessment Battery for Children, Second edition.
  The Bayley Scales of Infant and Toddler Development-Third Edition is an individually administered test designed to assess developmental functioning of infants and toddlers. The Bayley-III assesses development in five areas: cognitive, language, motor, social-emotional, and adaptive behavior.
  The Kaufman Assessment Battery for Children (K-ABC) is a clinical instrument for assessing cognitive development.
Time Frame: Week 24
Measure: Median (Full Range); unit: Months
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Months | -1.0 [-4 to 1] | -3.0 [-6 to 6]

19. Secondary Outcome: Change From Baseline in Age-equivalence Score as Assessed by VABS-II
Description: The age equivalent score represent the age in months of the typical and normal individual who would achieve the same result as the one who was tested.
  The age equivalent scores are assessed by Vineland™ Adaptive Behavior Scales, Expanded Interview Form, Second edition (VABS-II). The Vineland is designed to measure adaptive behavior of individuals from birth to age 90.
  The Vineland-II contains 5 domains each with 2-3 subdomains. The main domains are: Communication, Daily Living Skills, Socialization, Motor Skills, and Maladaptive Behavior.
Time Frame: Week 24
Measure: Median (Full Range); unit: Months
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Months | 1.0 [-9 to 2] | 0.0 [-3 to 24]

20. Secondary Outcome: Change From Baseline in Gray Matter Volume
Description: Grey matter contains most of the brain's neuronal cell bodies. The grey matter includes regions of the brain involved in muscle control, and sensory perception such as seeing and hearing, memory, emotions, speech, decision making, and self-control. The gray matter volume will be measured by volumetric magnetic resonance imaging (MRI).
Time Frame: Week 24
Measure: Median (Full Range); unit: mL
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
mL | 10.858 [-6.22 to 42.27] | 39.129 [-33.28 to 111.53]

21. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory (PedsQL™) Total Score
Description: Pediatric Quality of Life Inventory (PedsQL™) is a modular approach to measuring health-related quality of life (HRQOL) in healthy children and adolescents and those with acute and chronic health conditions. Lower scores indicate better functioning. Min score = 0, and max score = 144.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 3
Units on a scale | -9.3 (15.52) | -7.3 (14.9)

22. Secondary Outcome: Change From Baseline in PedsQL™ Family Impact Module Total Score
Description: Pediatric Quality of Life Inventory (PedsQL™) is a modular approach to measuring health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. The measure includes a scale, from where the categorical score "4", "3", "2", "1", and "0" was reversed and linearly transformed to a 0-100 scale to 4=0, 3=25, 2=50, 1=75 and 0=100, where 100 = minimum and 0 = maximum. The Total Score is the sum of all 36 items in the test divided by the number of items answered. Higher scores indicate better functioning.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Dose Group 1 | Dose Group 2
Number analyzed (Participants) | 3 | 2
Units on a scale | -9.77 (19.05) | 1.3 (3.11)

ADVERSE EVENTS:
Time Frame: The period for recording adverse events, including Serious Adverse Events (SAEs), began upon receiving the first dose of SOBI003 and ended at completion of the week 24 visit. In addition SAEs was reported from the time for signing the informed consent form until 28 days past the last dose of SOBI003.
Arm/Group | Dose Group 1 | Dose Group 2
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Group 1 (N=3) | Dose Group 2 (N=3)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Device related infestations (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Group 1 (N=3) | Dose Group 2 (N=3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (13) | 3 (15)
Vomiting (Gastrointestinal disorders) | 1 (2) | 3 (10)
Medical device site haemorrhage (General disorders) | 1 (1) | 0
Conjunctivitis (Infections and infestations) | 1 (1) | 0
Gastroenteritis (Infections and infestations) | 1 (2) | 0
Upper respiratory tract infection (Infections and infestations) | 3 (7) | 2 (3)
Viral infection (Infections and infestations) | 1 (1) | 0
Vascular access site occlusion (Injury, poisoning and procedural complications) | 1 (4) | 2 (5)
Tremor (Nervous system disorders) | 1 (1) | 2 (4)
Device damage (Product Issues) | 1 (2) | 0
Device malfunction (Product Issues) | 1 (1) | 0
Anxiety (Psychiatric disorders) | 1 (1) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (13)
Hyperaemia (Vascular disorders) | 1 (1) | 0
Aortic valve thickening (Cardiac disorders) | 0 | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 (1)
Abnormal faeces (Gastrointestinal disorders) | 0 | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 (6)
Faeces discoloured (Gastrointestinal disorders) | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | 0 | 1 (1)
Application site irritation (General disorders) | 0 | 1 (1)
Pyrexia (General disorders) | 0 | 3 (5)
Otitis media acute (Infections and infestations) | 0 | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 | 1 (2)
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 (3)
Blood fibrinogen increased (Investigations) | 0 | 1 (2)
Blood pressure diastolic increased (Investigations) | 0 | 1 (1)
Blood pressure systolic increased (Investigations) | 0 | 1 (1)
C-reactive protein increased (Investigations) | 0 | 1 (2)
CSF glucose decreased (Investigations) | 0 | 1 (1)
CSF protein increased (Investigations) | 0 | 1 (1)
Eosinophil count increased (Investigations) | 0 | 1 (2)
Haemoglobin increased (Investigations) | 0 | 1 (1)
Monocyte count decreased (Investigations) | 0 | 1 (1)
Neutrophil count increased (Investigations) | 0 | 1 (1)
Oxygen saturation decreased (Investigations) | 0 | 1 (5)
Platelet count decreased (Investigations) | 0 | 1 (1)
Red blood cell count increased (Investigations) | 0 | 1 (1)
White blood cell count increased (Investigations) | 0 | 1 (2)
Clonus (Nervous system disorders) | 0 | 1 (1)
Device dislocation (Product Issues) | 0 | 1 (1)
Restlessness (Psychiatric disorders) | 0 | 2 (3)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Vascular device user (Social circumstances) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT03423186/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-24): https://cdn.clinicaltrials.gov/large-docs/86/NCT03423186/SAP_001.pdf